CLINICAL TRIAL: NCT04823221
Title: A Real World Study to Evaluate the Feasibility, Preliminary Safety and Performance of Rezūm System in BPH Treatment in China (Rezūm RWS Study)
Brief Title: To Evaluate the Feasibility, Preliminary Safety and Performance of Rezūm System in BPH Treatment in China
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: U0719
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Results first posted 2022-02-17 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-03

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Rezūm system: The basic principle of the Rezūm System is to deliver a controlled amount of sterile water vapor directly into the hyperplastic tissue in the transition zone of the prostate using a transurethral approach .The stored thermal energy in the vapor is transferred directly onto the cell membranes as the vapor condenses and releases the heat of condensation, causing cell death. Inaddition, this thermal energy transfer collapses the vasculature within the treatment zone, resulting in a bloodless procedure. During procedure the water vapor is created by a heating element in the Rezūm Delivery Device,Saline flush during vapor delivery protects and preserves the urethra.
  Interventions: Device: Rezūm System

INTERVENTIONS:
Device: Rezūm System — The basic principle of the Rezūm System is to deliver a controlled amount of sterile water vapor directly into the hyperplastic tissue in the transition zone of the prostate using a transurethral approach .The stored thermal energy in the vapor is transferred directly onto the cell membranes as the vapor condenses and releases the heat of condensation, causing cell death. Inaddition, this thermal energy transfer collapses the vasculature within the treatment zone, resulting in a bloodless procedure. During procedure the water vapor is created by a heating element in the Rezūm Delivery Device,Saline flush during vapor delivery protects and preserves the urethra.

SUMMARY:
A real world study to evaluate the feasibility, preliminary safety and performance of Rezūm system in BPH treatment in China Rezūm RWS study

DETAILED DESCRIPTION:
This RWS study is to evaluate the feasibility, preliminary safety and performance of Rezūm system in BPH treatment in China, to generate local real world data from a Chinese BPH population.

The Rezūm System is intended to relieve symptoms, obstructions, and reduce prostate tissue associated with BPH. It is indicated for men ≥50 years of age with a prostate volume ≥ 30cm3 and ≤80cm3. The Rezūm System is also indicated for treatment of prostate with hyperplasia of the central zone and/or a median lobe.

ELIGIBILITY:
Inclusion Criteria:

* The subjects will provide written informed consent form and agree to data collection.
* The subjects who were diagnosed as BPH and treated by Rezūm procedure in Hainan medical pilot zone will be enrolled in this study.

Exclusion Criteria:

* This is a retrospective study without any formal exclusion criteria.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The Rezūm System is intended to relieve symptoms, obstructions, and reduce prostate tissue associated with BPH
Study Population: Up to 30 subjects who were diagnosed as BPH and treated with Rezūm system will be collected to get 22 treated subjects with valid data.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming Liu, Dr, Principal Investigator — Boao Yiling Life Care Center
Locations (1):
- Boao Yiling Life Care Center, Boao, Hainan, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rezūm System
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rezūm System
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 6
Age, Continuous [Median (Standard Deviation); unit: years] | 61 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 22
Weight [Median (Standard Deviation); unit: Kg] | 76.3 (9)
Prostate Volume (cm^3) [Median (Standard Deviation); unit: cm3]
  Doppler ultrasound(DUS) | 37.7 (9.5)
  Magnetic Resonance Imaging (MRI) | 43.7 (8.4)
Peak flow rate (Qmax)) [Median (Standard Deviation); unit: mL/second] | 11.9 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: International Prostate Symptom Score (IPSS) Change From Baseline to the Last Follow-up Date, Anywhere Between Month 3 - Month 6 Post Rezūm Procedure.
Description: International prostate symptom score (IPSS) is a questionnaire used to indicate the severity of LUTS symptoms, There are 7 questions relating to different symptoms subjects be experiencing.
  7 questions about patients' urinating include Incomplete emptying, Frequency, Intermittency, Urgency, Weak stream, Straining and Nocturia, every question have 0-5 scores according to Prostate Symptom, the higher score mean patient have more severe the symptoms.
  IPSS total score: the minimum score is 0 and maximum score are 35. IPSS total 0-7 scores are mild symptoms, IPSS total 8-19 scores are moderate symptoms and IPSS total 20-35 scores are severe symptoms The change was the value at the baseline minus the value at last follow-up date, anywhere between month 3 - month 6 minus
Time Frame: from baseline to the last follow-up date, anywhere between month 3 - month 6 post Rezūm procedure
Measure: Median (Standard Deviation); unit: scores on a scale
Arm/Group | Rezūm System
Number analyzed (Participants) | 22
scores on a scale | 14.9 (4.4)

2. Primary Outcome: Device Related Serious Complications From Rezūm Procedure to the Last Follow-up Date, Anywhere Between Month 3 - Month 6 Post Rezūm Procedure.
Description: Composite device related serious complications for this endpoint are defined as:
  1. Device perforation of the rectum or GI tract;
  2. Device related formation of fistula between the rectum and urethra;
  3. De novo severe urinary retention lasting more than 21 consecutive days post treatment.
Time Frame: from Rezūm procedure to the last follow-up date, anywhere between month 3 - month 6 post Rezūm procedure.
Measure: Number; unit: adverse events
Arm/Group | Rezūm System
Number analyzed (Participants) | 22
adverse events | 0

3. Secondary Outcome: Rezūm Procedure Time
Description: Rezūm procedure time is refers to the urethral entry of the catheter by Rezūm and exit after the ablation of the catheter by Rezūm
Time Frame: During Rezūm procedure
Measure: Median (Standard Deviation); unit: Minutes
Arm/Group | Rezūm System
Number analyzed (Participants) | 22
Minutes | 3.9 (1.6)

4. Secondary Outcome: Length of Catheterization
Description: Length of Catheterization is the date from date of catheter implantation to date of catheter removal
Time Frame: 1 month post Rezum procedure
Measure: Median (Standard Deviation); unit: days
Arm/Group | Rezūm System
Number analyzed (Participants) | 22
days | 4.8 (1.1)

5. Secondary Outcome: The Change of Peak Flow Rate (Qmax) From Baseline to the Last Follow-up Date, Anywhere Between Month 3 - Month 6 Post Rezūm Procedure.
Description: The change of Peak Flow Rate (Qmax) from baseline to the last follow-up date, anywhere between month 3 - month 6 post Rezūm procedure. Which are the value at the last follow-up date, anywhere between month 3 - month 6 minus value at baseline
Time Frame: from baseline to the last follow-up date, anywhere between month 3 - month 6 post Rezūm procedure.
Population: Only 11 subjects completed Qmax in 3-6 months
Measure: Median (Standard Deviation); unit: mL/second
Arm/Group | Rezūm System
Number analyzed (Participants) | 11
mL/second | 13.3 (9.9)

6. Secondary Outcome: Post Void Residual Urine Volume (PVR）
Description: The change of Post Void Residual Urine Volume (PVR）from baseline to the last follow-up date, anywhere between month 3 - month 6 post Rezūm procedure. The change are the baseline value minus the value at the last follow-up date, anywhere between month 3 - month 6 minus.
Time Frame: from baseline to the last follow-up date, anywhere between month 3 - month 6 post Rezūm procedure.
Population: Only 15 subjects completed PVR test in 3-6 month.
Measure: Median (Standard Deviation); unit: ml
Arm/Group | Rezūm System
Number analyzed (Participants) | 15
ml | 11.6 (22.4)

7. Secondary Outcome: Quality of Life (Qol)
Description: The change of Quality of Life from baseline to the last follow-up date, anywhere between month 3 - month 6 post Rezum procedure. There is only 1 question about Quality of life due to urinary symptoms which is 'If you were to spend the rest of your life with your urinary condition the way it is now, how would you feel about that?' This question have 0-6 scores according to patient's satisfaction about Quality of Life, the higher score mean patient have poor satisfaction.
  The change was the baseline value minus the value at the last follow-up date, anywhere between month 3 - month 6.
Time Frame: from baseline to the last follow-up date, anywhere between month 3 - month 6 post Rezum procedure
Population: Only 20 subjects completed Quality of Life testing in 3-6 months post Rezum procedure.
Measure: Median (Standard Deviation); unit: scores on a scale
Arm/Group | Rezūm System
Number analyzed (Participants) | 20
scores on a scale | 2.5 (0.9)

8. Secondary Outcome: Ejective Function (MSHQ-EjD)
Description: The change of Ejective function-Male Sexual Health Questionnaire Short Form- Ejaculation dysfunction（MSHQ-EjD ) from baseline to the last follow-up date, anywhere between month 3 - month 6 post Rezum procedure. Ejective function (MSHQ-EjD) is a questionnaire used to assess the ejective function. There are 4 questions relating to Ejaculation dysfunction which need patients to answer.
  3 questions about patients' ejective function assessing include completion of ejaculation, Strength of ejaculation and Volume of semen when ejaculation. Every question have 0-5 scores according to assessing the ejective function, the lower score mean patient have more severe the ejective function.
  MSHQ-EjD total score: the minimum score is 0 and maximum score are 15. The change are the value at the last follow-up date, anywhere between month 3 - month 6 minus value at baseline
Time Frame: from baseline to the last follow-up date, anywhere between month 3 - month 6 post Rezum procedure
Population: Only 18 subjects completed Ejective function assessment
Measure: Median (Standard Deviation); unit: scores on a scale
Arm/Group | Rezūm System
Number analyzed (Participants) | 18
scores on a scale | 2.6 (3.5)

9. Secondary Outcome: The Change of International Index of Erectile Function(IIEF) From Baseline to the Last Follow-up Date, Anywhere Between Month 3 - Month 6
Description: The change of the International Index of Erectile Function(IIEF) from baseline to the last follow-up date, anywhere between month 3 - month 6 post Rezum procedure. Erectile Function(IIEF) is a questionnaire used to assess the Sexual Health Inventory of men. There are 5 questions relating to Erectile Function which need patients to answer. Every question have 0-5 scores, the lower score mean patient have more severe the Erectile Function.
  The IIEF-5 is administered as a screening instrument for the presence & severity of ED in conjunction with the clinical assessment. The score is the sun of the responses to the five items, so that overall score may range from 0 to 25. A score of 20 or higher indicates a normal degree of erectile functioning. Low scores (10 or less) indicate moderate to severe ED.
  The change are the value at the last follow-up date, anywhere between month 3 - month 6 minus value at baseline
Time Frame: From baseline to the last follow-up date, anywhere between month 3 - month 6
Measure: Median (Standard Deviation); unit: scores on a scale
Arm/Group | Rezūm System
Number analyzed (Participants) | 18
scores on a scale | 2.7 (5.1)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected in 6 months post Rezūm procedure
Arm/Group | Rezūm System
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 22/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rezūm System (N=22)
Urethral disorder (Renal and urinary disorders) | 19 (19)
Haematuria (Renal and urinary disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT04823221/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT04823221/SAP_001.pdf